CLINICAL TRIAL: NCT04406155
Title: Bowel Preparation Before Three-dimensional Rectal Water Contrast Transvaginal Ultrasonography for Diagnosing the Presence and Describing the Characteristics of Rectosigmoid Endometriosis
Brief Title: Bowel Preparation Before 3D Rectal Water Contrast Transvaginal Ultrasonography for Rectosigmoid Endometriosis
Status: Completed | Type: Observational
Sponsor: Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia (Other)
Responsible Party: Principal Investigator, Simone Ferrero, Principal Investigator, Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia
Other Study IDs: BP-3DRWC-TVS-RECTOSIG
Record Dates: First submitted 2020-05-25; First posted 2020-05-28 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Endometriosis, Rectum
Keywords: rectosigmoid endometriosis; bowel preparation
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspicion of rectosigmoid endometriosis
  Interventions: Procedure: 3D-RWC-TVS with bowel preparation; Procedure: 3D-RWC-TVS without bowel preparation

INTERVENTIONS:
Procedure: 3D-RWC-TVS with bowel preparation — Rectal water contrast transvaginal ultrasonography is based on the distention of rectosigmoid with saline solution. Three-dimensional reconstructions convert standard 2D grayscale ultrasound acquisitions into a volumetric dataset.
  Bowel preparation is based on a low-residue diet given in the two days before the examination and a rectal enema administered a few hours before the procedure.
Procedure: 3D-RWC-TVS without bowel preparation — Rectal water contrast transvaginal ultrasonography is based on the distention of rectosigmoid with saline solution. Three-dimensional reconstructions convert standard 2D grayscale ultrasound acquisitions into a volumetric dataset.

SUMMARY:
Three-dimensional (3D) rendering may be employed during transvaginal rectal water-contrast transvaginal ultrasonography (RWC-TVS) for detecting the presence and describe the characteristics of rectosigmoid endometriosis. This study aims to evaluate the impact of bowel preparation on the diagnostic parameters of 3D-RWC-TVS in women with suspicion of rectosigmoid endometriosis.

DETAILED DESCRIPTION:
An accurate diagnosis of the presence, location and extent of the rectosigmoid endometriosis is of paramount importance for the clinicians in order to inform the patients on the potential surgical or medical treatments. It is well established that transvaginal ultrasonography is the first-line investigation in patients with suspicion of deep infiltrating endometriosis. An improvement in the performance of transvaginal ultrasonography in diagnosing rectosigmoid endometriosis may be obtained by using rectal water contrast during transvaginal ultrasonographic scan. In the last years, three-dimensional (3D) rendering has been employed during transvaginal ultrasound for benign gynecological diseases.

ELIGIBILITY:
Inclusion Criteria:

- pain and intestinal symptoms suggestive of rectosigmoid endometriosis

Exclusion Criteria:

* previous surgical diagnosis of intestinal endometriosis
* previous radiological diagnosis of intestinal endometriosis (based on Magnetic Resonance or double-contrast barium enema
* history of colorectal surgery (except appendectomy)
* contraindications to bowel preparation or computed colonography (such as non-- compliant patients and rectal malformations)
* previous bilateral ovariectomy
* psychiatric disorders

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with suspicion of rectosigmoid endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
To compare the accuracy of 3D-RWC-TVS with and without bowel preparation in the diagnosis of rectosigmoid endometriosis. | At maximum 6 months before laparoscopic surgical approach
  The results of imaging will be compared with surgical and histological findings.

SECONDARY OUTCOMES:
To compare the precision of 3D-RWC-TVS with and without bowel preparation in estimating the length (mid-sagittal diameter) of the rectosigmoid endometriotic nodules | At maximum 6 months before laparoscopic surgical approach
  The results of imaging will be compared with surgical and histological findings.
To compare the accuracy of 3D-RWC-TVS with and without bowel preparation in the diagnosis of multifocal rectosigmoid endometriosis. | At maximum 6 months before laparoscopic surgical approach
  The results of imaging will be compared with surgical and histological findings.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ferrero, MD, PhD, Study Director — IRRCS Ospedale Policlinico San Martino
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferrero S, Barra F, Stabilini C, Vellone VG, Leone Roberti Maggiore U, Scala C. Does Bowel Preparation Improve the Performance of Rectal Water Contrast Transvaginal Ultrasonography in Diagnosing Rectosigmoid Endometriosis? J Ultrasound Med. 2019 Apr;38(4):1017-1025. doi: 10.1002/jum.14790. Epub 2018 Sep 24. PMID 30246880
- [Background] Ferrero S, Scala C, Stabilini C, Vellone VG, Barra F, Leone Roberti Maggiore U. Transvaginal sonography with vs without bowel preparation in diagnosis of rectosigmoid endometriosis: prospective study. Ultrasound Obstet Gynecol. 2019 Mar;53(3):402-409. doi: 10.1002/uog.19194. Epub 2019 Feb 6. PMID 30079504